CLINICAL TRIAL: NCT03150290
Title: Energy Expenditure and Brown Adipose Tissue in Amyotrophic Lateral Sclerosis
Brief Title: Brown Adipose Tissue in ALS
Acronym: BATALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: C16-83; 2016-A01790-51 (Registry Identifier: RCB)
Record Dates: First submitted 2017-05-09; First posted 2017-05-12 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALS patients without weight loss. (Other): 18-FDG-PET. Indirect Calorimetry.
  Interventions: Other: Indirect Calorimetry.; Device: 18-FDG-PET
- ALS patients with weight loss. (Other): 18-FDG-PET. Indirect Calorimetry.
  Interventions: Other: Indirect Calorimetry.; Device: 18-FDG-PET

INTERVENTIONS:
Other: Indirect Calorimetry. — REE measurement
Device: 18-FDG-PET — 18-FDG-PET

SUMMARY:
Weight loss is a common phenomenon in ALS. During the course of the disease, difficulty in swallowing and mastication can be responsible for a decrease in caloric intake and thus for weight loss. However, significant weight loss can also be observed in patients with no feeding difficulties. About half of ALS patients have an increase in their resting energy consumption, but the origin of this "hypermetabolism" remains unknown. "Brown" fat is specialized in the production of heat. Unlike "white" fat that stores excess caloric intakes, brown fat consumes energy. In humans, brown fat has long been considered as absent in adults. However, recent imaging techniques have been able to detect brown fat deposits in some adult subjects. The aim of this study is thus to determine the role of brown fat on energy consumption in Amyotrophic Lateral Sclerosis.

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a progressive neurodegenerative disorder involving motor neurons of the cerebral cortex, brain stem and spinal cord. Motor neuron loss results in rapidly progressive muscle paralysis, usually leading to death from respiratory failure in 3-5 years.

Weight loss is a frequent phenomenon and an independent negative prognostic factor for survival in ALS. Involvement of bulbar muscles with dysphagia is likely to lead to decrease in energy intake resulting in negative energy balance. However, weight loss also occurs in non-dysphagic patients, and is not restricted to reduction in skeletal muscle mass but also involves fat mass reduction.

Hypermetabolism (i.e. elevation of resting energy expenditure, REE) have been reported in ALS in about 50% of ALS patients but the origin of this hypermetabolism remains unknown. Increase of REE seems paradoxical in the context of ALS because skeletal muscle mass, which accounts for a large proportion of energy consumption and heat production, is decreased in ALS patients. Brown adipose tissue (BAT) is another important organ for basal and inducible energy expenditure and thermogenesis. In humans, BAT is primarily found in infants and young children, and healthy adults has long been considered as almost devoid of functional BAT. However, a recent study using 18F-fluorodeoxyglucose (18F-FDG) positron-emission tomographic (PET) scan showed that depots of functional BAT were present in about 5% of adult humans, most commonly localized in the cervical-supraclavicular region. In an autopsy series, depots of BAT in the periadrenal region were found in 19/20 ALS patients. It has been estimated that, if present, 50 g of maximally stimulated brown tissue could represent up to 20% of REE expenditure in an adult human. The presence of substantial, functional, depots of BAT could thus participate in the increase of REE observed in ALS patients.

The primary objective of this study is to identify and quantify potential depots of functional BAT in ALS patients. Secondary objectives will be to correlate amount of detectable BAT with measured REE, clinical parameters evaluating ALS progression and biological parameters.

This study will include 5 patients referred to the Paris ALS center with a diagnosis of ALS and "unexplained" (i.e. not explained by severe dysphagia) loss of 5 percent or more of normal body weight in the last 6 months. 5 ALS patients without significant weight loss will also be included in the study as controls.

For each patient, measurement of REE will be performed by indirect calorimetry. The volume and activity of BAT will be determined using 18F-FDG PET whole body scans. Data on concomitant and past disorders (including cancer and diabete mellitus), smoking history, medication use, height, current and normal body weight, age and site of onset of ALS symptoms will be recorded. Functional motor impairment will be assessed using manual muscle testing and the revised ALS Functional Rating Scale as in routine clinical practice.

This study will be the first to investigate, using non-invasive procedures, the role of depots of functional BAT in ALS patients' metabolic dysfunction. The results will provide new insights on the origin and consequences of the dysregulation of metabolic homeostasis in ALS.

ELIGIBILITY:
10 ALS patients, fulfilling the following inclusion criteria:

* Aged 18 to 85 (inclusive)
* Possible, probable (clinically or laboratory) or definite ALS according to the revised version of the El Escorial World Federation of Neurology criteria
* With unexplained significant loss of weight of 5 percent (or more) of normal body weight in the last 6 months (n=5 subjects) Or - without weight loss (n= 5 subjects)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Quantification of depots of functional brown adipose tissue in ALS patients (grams) | performed at the first visit (1 day)
  measured by 18F-FDG-PET

CONTACTS AND LOCATIONS:
Locations (1):
- Paris Als Center, Salpetriere Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: No